CLINICAL TRIAL: NCT00020267
Title: Phase I Randomized Study of MAGE-12 Peptide Vaccine in Patients With Refractory Metastatic Cancer Expressing MAGE-12 Antigen
Brief Title: Vaccine Therapy in Treating Patients With Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068173; NCI-00-C-0182; NCI-1034; NCT00006074 (obsolete NCT alias)
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer; Adult Soft Tissue Sarcoma; Colorectal Cancer; Bone Cancer; Ovarian Sarcoma; Melanoma; Colon Cancer; Rectal Cancer; Breast Cancer; Eye Cancer; Uterine Sarcoma
Keywords: Ewing's family of tumors; adult soft tissue sarcoma; adult solid tumor; body system/site cancer; bone cancer; breast cancer; cancer; childhood cancer; childhood solid tumor; ciliary body and choroid melanoma, medium/large size; colon cancer; colorectal cancer; extraocular extension melanoma; eye cancer; female reproductive cancer; gastrointestinal cancer; genetic condition; intraocular melanoma; lung cancer; male breast cancer; melanoma; metastatic osteosarcoma; metastatic tumors of the Ewing's family; muscle cancer; musculoskeletal cancer; non-small cell lung cancer; osteosarcoma; osteosarcoma/malignant fibrous histiocytoma of bone; ovarian sarcoma; rectal cancer; recurrent adult soft tissue sarcoma; recurrent breast cancer; recurrent colon cancer; recurrent intraocular melanoma; recurrent melanoma; recurrent non-small cell lung cancer; recurrent osteosarcoma; recurrent rectal cancer; recurrent tumors of the Ewing's family; recurrent uterine sarcoma; skin tumor; solid tumor; stage IIIB, IV, recurrent, and metastatic breast cancer; stage IV adult soft tissue sarcoma; stage IV breast cancer; stage IV colon cancer; stage IV melanoma; stage IV non-small cell lung cancer; stage IV rectal cancer; stage IV uterine sarcoma; stage IVA adult soft tissue sarcoma; stage IVB adult soft tissue sarcoma; stage, Ewing's family of tumors; stage, adult soft tissue sarcoma; stage, breast cancer; stage, colon cancer; stage, intraocular melanoma; stage, melanoma; stage, non-small cell lung cancer; stage, osteosarcoma; stage, rectal cancer; stage, uterine sarcoma; thorax/respiratory cancer; uterine sarcoma
MeSH Terms: conditions — Lung Neoplasms; Sarcoma; Colorectal Neoplasms; Bone Neoplasms; Melanoma; Colonic Neoplasms; Rectal Neoplasms; Breast Neoplasms; Eye Neoplasms; Neuroectodermal Tumors, Primitive, Peripheral; Neoplasms; Uveal Melanoma; Gastrointestinal Neoplasms; Genetic Diseases, Inborn; Breast Neoplasms, Male; Osteosarcoma; Muscle Neoplasms; Carcinoma, Non-Small-Cell Lung; Histiocytoma, Malignant Fibrous; Skin Neoplasms; Recurrence | interventions — Interleukin-2; montanide ISA 51

INTERVENTIONS:
Drug: interleukin-2
Drug: MAGE-12 peptide vaccine
Drug: Montanide ISA-51

SUMMARY:
RATIONALE: Vaccines made from a peptide may make the body build an immune response and kill tumor cells.

PURPOSE: Randomized phase I trial to study the effectiveness of vaccine therapy in treating patients who have metastatic cancer that has not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity profile of MAGE-12 peptide vaccine in patients with refractory metastatic cancer that expresses MAGE-12 antigen.

II. Determine whether an immunologic response, as measured by an in vitro sensitization assay, can be obtained after administration of this regimen in these patients.

III. Determine a frequency of administration for this regimen based on immunologic response in these patients.

IV. Determine other immunologic parameters in these patients treated with this regimen.

V. Determine the clinical response rate in these patients treated with this regimen.

PROTOCOL OUTLINE: This is a randomized study. Patients are stratified according to disease (metastatic cutaneous melanoma vs other tumor types). Patients are randomized to one of two treatment arms.

Arm I: Patients receive MAGE-12 peptide vaccine emulsified in Montanide ISA-51 adjuvant subcutaneously (SC) weekly for 4 doses.

Arm II: Patients receive MAGE-12 peptide vaccine emulsified in Montanide ISA-51 adjuvant SC once every 3 weeks for 4 doses.

Patients with progressive disease may receive interleukin-2 IV over 15 minutes every 8 hours, beginning on the day after each immunization and continuing for up to 4 days. Patients achieving stable disease or a mixed, partial, or complete response continue on vaccine therapy alone for up to 24 total doses.

Patients are followed at 3 weeks.

PROJECTED ACCRUAL:

A total of 26-56 patients (13-28 per treatment arm) will be accrued for this study within 1 year.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Histologically documented metastatic cancer of one of the following types: Cutaneous melanoma Ocular melanoma Colorectal carcinoma Non-small cell lung cancer Breast carcinoma Sarcoma HLA-Cw*0702 positive MAGE-12 expression by RT-PCR amplified tissue analysis Failed prior standard therapy Measurable or evaluable disease No renal carcinoma Hormone receptor status: Not specified --Prior/Concurrent Therapy-- Biologic therapy: At least 3 weeks since prior biologic therapy for cancer No other concurrent biologic therapy for cancer Chemotherapy: At least 3 weeks since prior chemotherapy for cancer and recovered No concurrent chemotherapy for cancer Endocrine therapy: At least 3 weeks since prior hormonal therapy for cancer No concurrent hormonal therapy for cancer No concurrent steroids Radiotherapy: At least 3 weeks since prior radiotherapy for cancer and recovered No concurrent radiotherapy for cancer Surgery: Prior surgery for cancer allowed --Patient Characteristics-- Age: 16 and over Sex: Male or female Menopausal status: Not specified Performance status: ECOG 0-2 Life expectancy: Greater than 3 months Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 90,000/mm3 Hepatic: Bilirubin no greater than 1.6 mg/dL AST/ALT less than 3 times normal Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No cardiac ischemia, myocardial infarction, or cardiac arrhythmias (if receiving interleukin-2 (IL-2) therapy) Pulmonary: No obstructive or restrictive pulmonary disease (if receiving IL-2 therapy) Other: Not pregnant Negative pregnancy test Fertile patients must use effective contraception No active systemic infections No autoimmune disease, known immunodeficiency disease, or active primary or secondary immunodeficiency Hepatitis B surface antigen negative HIV negative No other active major medical illnesses (if receiving IL-2 therapy)

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-07

CONTACTS AND LOCATIONS:
Overall Officials: Francesco M. Marincola, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Surgery Branch, Bethesda, Maryland, United States